CLINICAL TRIAL: NCT06154135
Title: Insulin Delivery Using the DBLG1 Closed-loop Algorithm on Glycemic Control and Patient-reported Outcomes in Adults Living With Type 1 Diabetes: a Multicenter Real-world Observational Study in Belgium
Brief Title: Insulin Delivery Using the DBLG1 Closed-loop on Glycemic Control and PROMs in Adults Living With Type 1 Diabetes
Acronym: INLOOP
Status: Enrolling by invitation | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2022123
Record Dates: First submitted 2023-11-06; First posted 2023-12-01 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the impact of the DBLG1 hybrid closed-loop system on glycemic control and patient-reported outcomes in adults living with type 1 diabetes under real-life conditions.

DETAILED DESCRIPTION:
This is a multicenter real-world observational study analyzing data on the use of the DBLG1 system in patients with T1D treated in the participating centers in Belgium. Data from patients with T1D who start(ed) with the DBLG1 between may-01 2022 up to and including August-01 2023 will be analyzed. Data will be collected during clinical routine follow-up from electronic medical records, questionnaires, standard of care laboratory tests and CGM-data. Baseline data from before start (up to -12 months) of the DBLG1 system and follow-up data at 4, 8, 12, 16, 20 and 24 months will be analyzed. There are no medical interventions, nor extra visits or laboratory tests planned outside normal clinical routine. Glycemic control and patient-reported outcomes during follow-up will be compared with glycemic control and patient-reported outcome data at baseline.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 diabetes
* aged 18 years and older
* starting with the DBLG1 system in the participating centers
* who signed the informed consent

Exclusion Criteria:

* patients who do not have type 1 diabetes
* younger than 18 years
* who do not start with the DBLG1 system
* who are not able to sign the informed consent
* who do not want to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T1D, aged 18 years and older, who start with the DBLG1 system in Belgium
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Time in range | 12 months after start
  Change in the percentage of time spent in range (sensor glucose 70-180 mg/dL) from before start to 12 months after start of the DBLG1 system

SECONDARY OUTCOMES:
Time in range [exc. primary outcome] | from before start to 4,8,12 and 24 months after start, with the exclusion of the primary outcome
  Change in the percentage of time spent in range (sensor glucose 70-180 mg/dL) after start of the DBLG1 system, with exclusion of the primary endpoint
Time in tigh range | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent in tigh range (sensor glucose 70-140 mg/dL) after start of the DBLG1 system.
Time in level 2 hypoglycemia | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent in level 2 hypoglycemia (sensor glucose below 54 mg/dL) after start of the DBLG1 system.
Time in level 1 hypoglycemia | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent in level 1 hypoglycemia (sensor glucose < 70 mg/dL and >=54 mg/dl) after start of the DBLG1 system.
Time below range | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent below range (sensor glucose < 70 mg/dL) after start of the DBLG1 system.
Time above range | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent above range (sensor glucose >180 mg/dL) after start of the DBLG1 system.
Time in level 2 hyperglycemia | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent in level 2 hyperglycemia (sensor glucose >250 mg/dL) after start of the DBLG1 system.
Time in level 1 hyperglycemia | from before start to 4,8,12 and 24 months after start
  Change in the percentage of time spent in level 1 hyperglycemia (sensor glucose >180 mg/dL and <= 250 mg/dl)) after start of the DBLG1 system.
Glycemic variability | from before start to 4,8,12 and 24 months after start
  Change in Coefficient of variation (CV) and standard deviation (SD) after start of the DBLG1 system.
Mean glucose concentration | from before start to 4,8,12 and 24 months after start
  Change in mean glucose concentration after start of the DBLG1 system.
HbA1c | from before start to 4,8,12 and 24 months after start
  Change in HbA1c (%) after start of the DBLG1 system.
Correlation between clinical characteristics and HbA1c changes | from before start to 4,8,12 and 24 months after start
  Correlation between recorded clinical characteristics and HbA1c changes after start of the DBLG1 system.
Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 | from before start to 4,8,12 and 24 months after start
  Change in Patient's Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire (scale: 0 (low quality of life) - 100 (high quality of life))
Clarke hypoglycemia awareness survey | from before start to 4,8,12 and 24 months after start
  Change in hypoglycemia awareness measured by the Clarke hypoglycemia awareness survey (scale: unaware (≥4 times "R" or once "U") or aware (<4 times "R"))
Gold scale | from before start to 4,8,12 and 24 months after start
  Change in hypoglycemia awareness measured by the Gold-scale (scale: 1 (aware) - 7 (unaware))
Hypoglycemia Fear Survey (HFS-II) | from before start to 4,8,12 and 24 months after start
  Change in fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry (scale: 0 (not worried) - 72 (very worried))
PAID-SF questionnaire | from before start to 4,8,12 and 24 months after start
  Change in distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire (scale: 0 (no distress) - 20 (very distressed))
Diabetes Impact and Device Satisfaction Scale (DIDSS) | from before start to 4,8,12 and 24 months after start
  Impact of diabetes and device satisfaction by the Diabetes Impact and Device Satisfaction Scale (scale: device satisfaction = 7 (not satisfied) - 70 (very satisfied); diabetes impact = 4 (low impact) - 40 (high impact))
Diabetes Treatment Satisfaction Questionnaire, Status (DTSQs) | from before start to 4,8,12 and 24 months after start
  Treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire, status (DTSQs. Scale: 0 (low satisfaction) - 36 (high satisfaction))
Reasons to stop using the DBLG-1 device | when the patient stops using the DBLG-1 system
  Self-developed questionnaire about the reasons the patient stopped using the DBLG-1 device (multiple choice)

OTHER OUTCOMES:
Composite endpoint of HbA1c and Time in Hypoglycemia | from before start to 4,8,12 and 24 months after start
  Composite endpoint of the percentage of participants reaching HbA1c <7% AND time in hypoglycemia (sensor glucose < 70 mg/dL) less than 4% of time after start of the DBLG1 system
Severe hypoglycemia | from before start to 4,8,12 and 24 months after start
  Change in Severe Hypoglycemia frequency after start of the DBLG1 system
Diabetic ketoacidosis | from before start to 4,8,12 and 24 months after start
  Change in diabetic ketoacidosis frequency after start of the DBLG1 system
Hospitals visits and/or admissions | from before start to 4,8,12 and 24 months after start
  Evolution of number of hospitals visits and/or admissions because of severe hypoglycemia or diabetic ketoacidosis from before start to 12 months after start of the DBLG1 system
Work and school absenteeism | from before start to 4,8,12 and 24 months after start
  Evolution of work and school absenteeism (number of days) after start of the DBLG1 system
Unplanned contacts with the diabetes team | from before start to 4,8,12 and 24 months after start
  Evolution of frequency of unplanned contacts with the diabetes team after start of the DBLG1 system
Change in body weight | from before start to 4,8,12 and 24 months after start
  Evolution of body weight (kg) after start of the DBLG1 system
Change in total daily dose of insulin | from before start to 4,8,12 and 24 months after start
  Evolution of total daily dose of insulin after start of the DBLG1 system
Indications for use of the DBLG-1 system (multiple options (non-ordinal)) | before start
  Indications for use of the DBLG-1 system measured by a self-developed questionnaire (multiple options (non-ordinal))
Patients who stop using the DBLG-1 system | from 4,8,12 and 24 months after start
  Number of patients who stop using the DBLG-1 system

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Crenier, PhD, Principal Investigator — CUB - Hôpital Erasme
Locations (12):
- Belgium (12):
  - Department of Endocrinology, OLVZ Aalst, Aalst
  - Department of Endocrinology, Imeldaziekenhuis, Bonheiden
  - Department of Endocrinology, ULB-Hôpital Erasme, Brussels
  - Department of Endocrinology and Nutrition, Cliniques Universitaires St. Luc, Brussels
  - Department of Endocrinology, UZ Antwerpen, Edegem
  - Department of Endocrinology and metabolic diseases, UZ Gent, Ghent
  - Department of Endocrino-Diabetology, Grand Hôpital de Charleroi - site Saint-Joseph, Gilly
  - Department of Endocrinology, UZ Leuven, Leuven
  - Department of Diabetes, Nutrition and Metabolic disorders, CHU de Liège - site du Sart Tilman, Liège
  - Department of Endocrinology, CHR de la Citadelle, Liège
  - Department of internal Medicine, CHU de Charleroi - Hôpital Civil Marie Curie, Lodelinsart
  - Department of Endocrinology, CHR Mons-Hainaut (Warquignies), Mons

IPD SHARING:
Plan to Share IPD: Yes
The protocol is published online
Supporting Information: Study Protocol
Time Frame: Available since May,1 2022
Access Criteria: open access
URL: https://www.inami.fgov.be/SiteCollectionDocuments/fiche_approuvement_tao_diabete_2.pdf